CLINICAL TRIAL: NCT00006475
Title: An Open-Label Study to Determine the Efficacy and Safety of STI571 in Patients With Chronic Myeloid Leukemia in Blast Crisis
Brief Title: STI571 in Treating Patients With Chronic Myelogenous Leukemia in Blast Crisis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068302; NOVARTIS-CSTI5710115
Record Dates: First submitted 2000-11-06; First posted 2004-04-26 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; Philadelphia chromosome negative chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: STI571 may interfere with the growth of cancer cells and may be an effective treatment for leukemia.

PURPOSE: Phase II trial to study the effectiveness of STI571 in treating patients who have chronic myelogenous leukemia in blast crisis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety profile of STI571 in patients with chronic myelogenous leukemia in blast crisis. II. Provide expanded access of this treatment to these patients. III. Determine the rate of hematological response and duration of response in patients treated with this regimen. IV. Determine the improvements in symptomatic parameters in patients treated with this regimen. V. Determine the cytogenetic response in patients treated with this regimen. VI. Determine the overall survival in patients treated with this regimen.

OUTLINE: This is an expanded-access, multicenter study. Patients receive oral STI571 daily. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients who are considered to have benefited may continue treatment beyond 1 year.

PROJECTED ACCRUAL: Not determined

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of chronic myelogenous leukemia (CML) in blast crisis, defined by at least one of the following: 30% blasts in peripheral blood and/or bone marrow Flow cytometry criteria Extramedullary disease other than spleen, lymph node, and/or liver involvement Newly diagnosed CML in blast crisis OR CML in blast crisis with prior therapy for accelerated or blastic phases Philadelphia (Ph) chromosome positive OR Ph chromosome negative and Bcr/Abl positive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: SGOT and SGPT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver involvement) Bilirubin no greater than 3 times ULN Renal: Creatinine no greater than 2 times ULN Cardiovascular: No grade 3 or 4 cardiac disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception during and for at least 2 weeks after study for women and for at least 3 months after study for men No history of noncompliance with medical regimens No serious concurrent medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 48 hours since prior interferon alfa At least 6 weeks since prior hematopoietic stem cell transplantation No concurrent anticancer biologic therapy Chemotherapy: At least 6 weeks since prior busulfan At least 24 hours since prior hydroxyurea At least 2 weeks since prior homoharringtonine At least 1 week since prior low-dose cytarabine (less than 30 mg/m2 every 12-24 hours daily) At least 2 weeks since prior moderate-dose cytarabine (100-200 mg/m2 for 5-7 days) At least 4 weeks since prior high-dose cytarabine (1-3 g/m2 every 12-24 hours for 6-12 doses) At least 3 weeks since prior anthracyclines, mitoxantrone, or etoposide No concurrent anticancer chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 4 weeks since other prior investigational agents No other concurrent anticancer investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Monteleone, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Corporation, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Hensley ML, van Hoomissen IC, Krahnke T, et al.: Imatinib in chronic myeloid leukemia (CML): outcomes in >7000 patients treated on expanded access program (EAP). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2328, 2003.
- [Result] van Hoomissen IC, Hensley ML, Krahnke T, et al.: Imatinib expanded access program (EAP): results of treatment in >7000 patients with chronic myeloid leukemia (CML). [Abstract] Blood 102 (11): A-3370, 2003.